CLINICAL TRIAL: NCT00730210
Title: Treatment of Hypoparathyroidism With Subcutaneous PTH (1-84) Injections: Effects on Muscle Function and Quality of Life
Acronym: HypoPTH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT #008-000606-36)
Record Dates: First submitted 2008-08-04; First posted 2008-08-08 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Hypoparathyroidism
Keywords: Hypoparathyroidism; HypoPTH; PTH
MeSH Terms: conditions — Hypoparathyroidism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- a: PTH (1-84) 100 ug s.c.inj. once a day (Active Comparator): PTH (1-84) 100 ug subcutaneous injections once a day
  Interventions: Drug: a: PTH (1-84)
- b: placebo 100 ug s.c. inj. once a day (Placebo Comparator): placebo 100 ug sub cutaneous injection once a day
  Interventions: Drug: b:placebo

INTERVENTIONS:
Drug: a: PTH (1-84) — preotact 100 microgram subcutaneous a day in 6 months
  Other Names: preotact
  Arms: a: PTH (1-84) 100 ug s.c.inj. once a day
Drug: b:placebo — 100 microgram placebo subcutaneous a day for 6 months
  Other Names: Placebo
  Arms: b: placebo 100 ug s.c. inj. once a day

SUMMARY:
The aim of the study is to assess whether PTH (1-84) therapy posses advantages compared to conventional treatment in patients with hypoparathyroidism on muscle function, quality of life, calcium homeostasis, bone metabolism, and body composition.

DETAILED DESCRIPTION:
Hypoparathyroidism is one of the only hormonal insufficiency states that is usually not treated by replacing the missing hormone. Currently, Standard therapy includes treatment with calcium and an 1alpha-hydroxylated forms of vitamin D (e.g. calcitriol or alphacalcidol) in order to relieve the symptoms associated with hypocalcaemia. However, recent studies have shown that calcium homeostasis can be well regulated by PTH replacement therapy in patients with hypoparathyroidism. It seems that PTH treatment is safe and that it even may posses advantages compared to conventional treatment with vitamin D. As the renal calcium excretion is decreased by PTH therapy, the risk of renal calcifications causing an impaired renal function may be reduced. In addition, some of the hypoparathyroid patients treated with PTH reported less fatigue and increased endurance in response to treatment. This may be due to either a better regulated (i.e. more physiological) calcium homeostasis during PTH therapy, or due to a direct effect of PTH on the neuromuscular system. Therefore, further studies are needed on the effects of PTH replacement in patients with hypoparathyroidism.

Outcome measures:

* Muscle- and balance function: Effects of treatment on muscle strength and balance function are determined using a dynamometer and a stadiometer (Meititur Ltd, Finland). In addition, effects of treatment on muscle function are assessed through muscle biopsies, electromyographic, echocardiography, and by biochemical measures (muscle enzymes).
* Quality of life: Effect of treatment on indices of quality of life is assessed using the SF-36v2- and the WHO-Five Well-Being Index (WHO-5)-survey.
* Calcium homeostasis, bone metabolism, and body composition. Effects of treatment are assessed by measurements of calcitropic hormones, biochemical markers of bone turnover, and iliac crest biopsies. In addition, bone mineral density and body composition is measured.

ELIGIBILITY:
Inclusion Criteria:

* A low endogenous PTH production as verified by low plasma levels of intact PTH, necessitating treatment with 1alpha-hydroxylated vitamin D analogs.
* At least one years of continuous alphacalcidol, calcitriol, or dihydrotachysterol treatment prior to study entry.
* Prior to start of study, participants are required to have received a daily supplement of at least 400 IU (10 microgram) of vitamin D (ergocalciferol or cholecalciferol) for at least 3 months or 25hydroxyvitamin D levels above 50 nmol/l. Subjects may be treated with ergocalciferol or cholecalciferol during a run-in period of three months before entering the study.
* Normal plasma magnesium level (If not, magnesium supplements may be provided during a 3 months run in period).
* Plasma calcium levels within the normal reference range or slightly below (P-Ca ionized 1.00 to 1.30).
* Use of safe contraceptive methods (fertile women).
* Speak and read Danish.

Exclusion Criteria:

* Known allergic reactions to any of the compounds in the trial medication.
* Severely impaired renal function (plasma creatinine > 200 micromol/l).
* Severely impaired hepatic function (Plasma alanine aminotransferase (ALAT) > 100 U/l and/or alkaline phosphatase > 400 U/l).
* Previous or present malignancies (except a treated skin cancer that is not melanoma or treated carcinoma in situ, 2 years since last therapy).
* Prior radiation therapy involving the skeleton.
* Current treatment with raloxifene, calcitonin, systemic corticosteroids above 5 mg a day, fluoride, lithium, PTH, or digoxin.
* Treatment with anticonvulsant's (within the last 2 years).
* Immobilization (more than two week within the last 6 months).
* Granulomatous disease.
* Paget's disease of bone.
* Pregnancy / planned within the next year. Hospitalized due to chronic drug or alcohol abuse. Severe malabsorption syndrome.
* Major medical or social problems that will be likely to preclude participation for one year.
* Unwillingness to participate.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2008-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Increase in maximal voluntary knee extension | 6 months

SECONDARY OUTCOMES:
Balance function: Is assessed using a stadiometer (Meititur Ltd, Finland) | 6 months
Effect of treatment on indices of quality of life is assessed using the SF-36v2- and WHO-Five Well-Being Index (WHO-5)-survey. | 6 months
Effects of treatment on muscle function are assessed through muscle biopsies, electromyographic, and by biochemical measures (muscle enzymes). | 6 months
Bone mineral density and body composition is measured | 6 months
Calcium homeostasis and bone metabolism. Effects of treatment are assessed by measurements of calcitropic hormones, biochemical markers of bone turnover, and bone biopsies | 6 months
Q CT scan of hip and spine | 6 months
Effects of treatment on diurnal variations of measured biochemical indices, as assessed at the end of the treatment period | 24 hours at the end of the 6 month treatment period
Effects of treatment on indices of cardiovascular health (ECG and blood pressure), as measured at the end of the treatment period just prior to and 1 hour after injection of study medication. | at the end of the 6 months treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Lars Rejnmark, MD,DrMed, Principal Investigator; Tanja Sikjær, MD, Principal Investigator
Locations (1):
- Osteoporoseklinikken, Aarhus University Hospital, Aarhus, Jutland, Denmark

REFERENCES:
- [Derived] Grunewald TA, Liebi M, Wittig NK, Johannes A, Sikjaer T, Rejnmark L, Gao Z, Rosenthal M, Guizar-Sicairos M, Birkedal H, Burghammer M. Mapping the 3D orientation of nanocrystals and nanostructures in human bone: Indications of novel structural features. Sci Adv. 2020 Jun 12;6(24):eaba4171. doi: 10.1126/sciadv.aba4171. eCollection 2020 Jun. PMID 32582855
- [Derived] Harslof T, Sikjaer T, Sorensen L, Pedersen SB, Mosekilde L, Langdahl BL, Rejnmark L. The Effect of Treatment With PTH on Undercarboxylated Osteocalcin and Energy Metabolism in Hypoparathyroidism. J Clin Endocrinol Metab. 2015 Jul;100(7):2758-62. doi: 10.1210/jc.2015-1477. Epub 2015 May 8. PMID 25955226
- [Derived] Sikjaer T, Rolighed L, Hess A, Fuglsang-Frederiksen A, Mosekilde L, Rejnmark L. Effects of PTH(1-84) therapy on muscle function and quality of life in hypoparathyroidism: results from a randomized controlled trial. Osteoporos Int. 2014 Jun;25(6):1717-26. doi: 10.1007/s00198-014-2677-6. Epub 2014 Apr 1. PMID 24687385